CLINICAL TRIAL: NCT02378350
Title: A Multicenter, Randomized, Open-Label Study of Quality of Life in Peritoneal Dialysis and Conventional In-Center Hemodialysis (ChinaQ Study)
Brief Title: Quality of Life on Peritoneal Dialysis Versus Hemodialysis in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8339-001
Record Dates: First submitted 2015-02-10; First posted 2015-03-04 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESRD patients receiving HD treatment (Active Comparator): no investigational drug involved. Only observe therapy treatment
  Interventions: Device: Hemodialysis treatment (no specific device is defined)
- ESRD patients receiving PD treatment (Experimental): no investigational drug involved. Only observe therapy treatment
  Interventions: Drug: Peritoneal Dialysis treatment (no specific drug is defined)

INTERVENTIONS:
Device: Hemodialysis treatment (no specific device is defined)
  Arms: ESRD patients receiving HD treatment
Drug: Peritoneal Dialysis treatment (no specific drug is defined)
  Arms: ESRD patients receiving PD treatment

SUMMARY:
This is a multicenter, randomized, open-label study to compare QoL in subjects with end-stage renal disease (ESRD) requiring PD or conventional in-center HD treatment.

Primary Objective: The primary objective is to demonstrate non-inferiority of peritoneal dialysis (PD) treatment as compared to hemodialysis (HD) treatment after approximately 1 year of therapy using the Kidney Disease Quality of Life-Short Form (KDQoL-SF) questionnaire domain of burden of kidney disease.

Secondary Objectives: The secondary objectives are to observe and summarize the following parameters in subjects receiving PD or HD treatment except for the remaining domains of QoL instrument KDQoL-SF™ (version 1.3) and the 2 individual QoL items scored as single items, which will be compared between the 2 treatment groups:

* Mortality rates
* Switch (PD to HD or HD to PD)
* Transplantation rate
* Cause of death
* Dialysis adequacy (ie, urea clearance time normalized by total body water, which is the volume of distribution of urea [Kt/V urea] to determine the proportion of subjects meeting standards of care for dialysis adequacy).
* 24-hour urine volume
* Change in hemoglobin and S-phosphate levels, and the percentages of subjects with values within the target range
* Change in serum albumin
* Frequency of adverse events (AEs) and serious AEs (SAEs), including abnormal laboratory test findings with clinical significance

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their legal representative who are able to understand and have voluntarily signed the informed consent form (ICF)
2. Male or female subjects aged 18 years or older at the time of randomization
3. Subjects diagnosed with ESRD (ie, an estimated glomerular filtration rate ≤15 mL/min/1.73 m2 body surface area) and who the Investigator anticipates will require maintenance dialysis therapy within 10 weeks after signing the ICF
4. Subjects who, as judged by the Investigator, are able to comprehend the standardized, predialysis education program and have completed this education prior to signing the ICF
5. Subjects or their legal representative who, as judged by the Investigator, are capable of being trained for home-based PD
6. Subjects who are able to adhere to the study visit schedule and other protocol requirements
7. Subjects who are able to come to HD clinics as required by the protocol
8. Subjects who, as judged by the Investigator, are expected to remain on dialysis for at least 48 weeks
9. Subjects who have normal liver function, as judged by the Investigator
10. Female subjects of childbearing potential must have negative serum or urine pregnancy test at Screening. Sexually active women of childbearing potential must agree to use adequate contraceptive methods, as judged by the Investigator, while in the study

Exclusion Criteria:

1. Subjects who are HIV positive
2. Subjects who have already received maintenance dialysis. Subjects are not excluded if a functional dialysis access is present ≤4 weeks before Screening for back-up purposes or for acute treatment of life-threatening uremic symptoms, electrolyte abnormalities or fluid overload
3. Subjects who have an active infection or other condition that the Investigator determines may jeopardize their ability to receive either modality of dialysis treatment or would preclude participation in the study
4. Subjects who report a history of illicit drug use or a regular or daily alcohol consumption of ≥4 alcoholic drinks per day in the 2 years before Screening
5. Subjects who have previously received renal transplantation and are currently prescribed immunosuppressive therapy
6. Subjects who are currently using any investigational drug
7. Subjects who are currently enrolled in other clinical studies
8. Subjects who are unwilling or unable to fully comply with the visits and assessments required by the protocol
9. Subjects who are not eligible for either PD or HD, as judged by the Investigator, due to:

   * Peritoneal dialysis: documented extensive intra-peritoneal adhesions or other conditions in which PD is contraindicated
   * Hemodialysis: severe cardiac instability or other conditions in which HD is contraindicated
10. Subjects who have a malignancy requiring chemotherapy or radiation therapy
11. Subjects undergoing temporary dialysis treatment between the Screening visit and Day 1 visit that is expected to exceed 6 weeks in duration
12. Subjects who have a life expectancy of < 48 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
1 year of therapy using the Kidney Disease Quality of Life-Short Form (KDQoL-SF) questionnaire | 1 year

SECONDARY OUTCOMES:
Mortality rates | 1 year
Switch (PD to HD or HD to PD) | 1 year
Transplantation rate | 1 year
Cause of death | 1 year
Dialysis adequacy | 1 year
24-hour urine volume | 1 year
Change in hemoglobin | 1 year
Change in serum albumin | 1 year
Frequency of adverse events (AEs) and serious AEs (SAEs), including abnormal laboratory test findings with clinical significance | 1 year
Change in S-phosphate levels | 1 year

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital , Sun Yet-Sen University, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The 2nd Shenzhen Municipal People's Hospital, Shenzhen, Guangdong
  - Guizhou Province People's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Traditional Chinese Medicine Hospital of Wuhan, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi province people's hospital, Nanchang, Jiangxi
  - Nanchang First Affiliated Hospital, Nanchang, Jiangxi
  - First Hospital of Affiliated of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Ningxia Medical University, Yingchuan, Ningxia
  - Renji Hospital , Shanghai Jiaotong University , School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai 455 Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Ethier I, Hayat A, Pei J, Hawley CM, Johnson DW, Francis RS, Wong G, Craig JC, Viecelli AK, Htay H, Ng S, Leibowitz S, Cho Y. Peritoneal dialysis versus haemodialysis for people commencing dialysis. Cochrane Database Syst Rev. 2024 Jun 20;6(6):CD013800. doi: 10.1002/14651858.CD013800.pub2. PMID 38899545